CLINICAL TRIAL: NCT02455999
Title: Dose-finding Study to Assess the Safety and Effect of SYL1001 in Patients With Ocular Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYL1001_III
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Ocular Pain; Dry Eye Syndrome
MeSH Terms: conditions — Eye Pain; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- SYL1001 eye drops dose C (Experimental): SYL1001 eye drops dose C administration via the ophthalmic route
  Interventions: Drug: SYL1001
- SYL1001 eye drops dose D (Experimental): SYL1001 eye drops dose D administration via the ophthalmic route
  Interventions: Drug: SYL1001
- Placebo (Placebo Comparator): Placebo eye drops administration via the ophthalmic route
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYL1001 — SYL1001 eye drops dose C administration for 10 consecutive days
  Arms: SYL1001 eye drops dose C
Drug: SYL1001 — SYL1001 eye drops dose D administration for 10 consecutive days
  Arms: SYL1001 eye drops dose D
Drug: Placebo — Placebo eye drops administration for 10 consecutive days
  Arms: Placebo

SUMMARY:
The aim of this pilot study is to compare the analgesic effect of two strengths of SYL1001 eye drops versus placebo in patients with ocular pain associated with Dry Eye Syndrome. General and local tolerability are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent to participate in the study, after having received all information relating to the design, aims and possible risks resulting therefrom.
* Common symptoms of persistent, daily, mild to moderate dry eye lasting more than three months: OSDI scale between 13-70 and VAS scale between 2 -7.
* Eye tests in both eyes: Corneal fluorescein staining (Oxford scale > 0), Tear break-up time < 10 seconds and Schirmer's test with anaesthesia < 10 mm/5min.

Exclusion criteria:

* Women who are pregnant or breastfeeding or who have a positive urine pregnancy test. Women who do not commit to use a medically acceptable method of contraception from the time of selection and throughout the study.
* Any current, relevant disease, including respiratory disease, cardiovascular disease, endocrine disease, neurological disease, haematological disease, kidney disease, oncological disease, liver disease, gastrointestinal dysfunction, hypertension or active acute infectious processes.
* Previous chronic or recurrent processes which, according to the investigator, could affect the development of the study.
* Concomitant use of other medications with analgesic activity by any route of administration at the time of entry into the study.
* Change in any concomitant eye and/or systemic medication of the patient one month before the study and during the study.
* Changes in the pre-established administration schedule of artificial tears during the 15 days before the study and during the 10 days of the study.
* Initiation of treatment with cyclosporine or changes in the dosage or administration schedule of cyclosporine within the 6 months before inclusion in the study.
* History of hypersensitivity to drugs.
* Use of contact lenses during the treatment and previous 15 days.
* History of drug abuse or drug or alcohol dependence.
* Laboratory abnormalities which, in the investigator's opinion, are clinically significant.
* Previous refractive surgery.
* Having participated in another clinical trial within the 2 months prior to inclusion.
* Another eye disease that is significant in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from the baseline scoring of eye pain on the Visual Analogue Scale (VAS) | 10 consecutive days
Change from the baseline scoring of ocular discomfort in the Ocular Surface Disease Index (OSDI) | 10 consecutive days
Change from the baseline scoring after fluorescein staining of the cornea | 10 consecutive days
Frequency of occurrence of conjunctival hyperaemia | 10 consecutive days

SECONDARY OUTCOMES:
Change from baseline in vital signs | 10 consecutive days
Change from baseline in standard laboratory parameters | 10 consecutive days
Assessment of Adverse Events (AEs) as a measure of SYL1001 safety | 20 consecutive days
Change from baseline in standard ocular parameters | 10 consecutive days

CONTACTS AND LOCATIONS:
Locations (6):
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Eye Clinic Dr. Krista Turman, Tallinn
- Spain (4):
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital U. Clínico San Carlos, Madrid
  - Clínica Universidad de Navarra, Pamplona

REFERENCES:
- [Derived] Benitez-Del-Castillo JM, Moreno-Montanes J, Jimenez-Alfaro I, Munoz-Negrete FJ, Turman K, Palumaa K, Sadaba B, Gonzalez MV, Ruz V, Vargas B, Paneda C, Martinez T, Bleau AM, Jimenez AI. Safety and Efficacy Clinical Trials for SYL1001, a Novel Short Interfering RNA for the Treatment of Dry Eye Disease. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6447-6454. doi: 10.1167/iovs.16-20303. PMID 27893109